CLINICAL TRIAL: NCT00615979
Title: Far Forward Battlefield Telemedicine:Ultrasound Guidance System (UGS)
Brief Title: Far Forward Battlefield Telemedicine: Evaluation of Handheld Ultrasound
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 5279; DAMD17-02-2-0040 (Other: USAMRMC)
Record Dates: First submitted 2007-12-26; First posted 2008-02-14 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Thoracic Injuries
Keywords: trauma; portable ultrasound; telemedicine; Department of Defense
MeSH Terms: conditions — Thoracic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Miniature echo machine: Diagnostic capabilities Wireless transfer
  Interventions: Device: Miniature echo machine

INTERVENTIONS:
Device: Miniature echo machine — Images captured and real-time and store-and-forward file transfers performed

SUMMARY:
The goal of this study is to improve survival of battlefield trauma through ultrasound telemedicine and remotely guided therapeutics.

DETAILED DESCRIPTION:
Specific aims to meet to improve the survival of battlefield trauma are 1)validation of portable ultrasound for diagnosis of various medical and surgical emergencies, ie cardiac tamponade, intraabdominal hemorrhage, 2)Extension of our expertise in digital echocardiography and local telemedicine to support other centers in such procedures as TEE 3)development of wireless telemedicine systems for rapid relay of ultrasonic images from portable ultrasound system to a remote review station. 4)development of a precision guide for diagnostic and therapeutic percutaneous procedures using ultrasound guidance 5)combining wireless telemetry with the guided percutaneous access tool to permit remotely guided emergency procedures 6)augmenting this work(2D/echo) with 3D/echo.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 yrs old
* Scheduled for clinical echocardiogram

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for clinical echocardiographic study Patients with possible diagnosis of cardiac tamponade
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2002-10 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Validation of small portable ultrasound units | single time point
  paired t-testing and linear regression will be used to test the hypothesis that the small system is equivalent to the full-featured one (mean difference in values not different from 0 and slope of the regression line not different

CONTACTS AND LOCATIONS:
Overall Officials: James Thomas, MD, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No